CLINICAL TRIAL: NCT02487147
Title: Evaluation of Free Air Portable Air Powered Respirator System for Prevention of Influenza Transmission
Brief Title: Evaluation of Free Air Portable Air Powered Respirator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Free Air (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00031388
Record Dates: First submitted 2015-06-26; First posted 2015-07-01 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2018-10

CONDITIONS: Influenza
Keywords: Live Attenuated Influenza Vaccine (FluMist); Free Air Portable Air Powered Respirator; N95 Respirator; Personal Protective Equipment; Viral Transmission
MeSH Terms: conditions — Influenza, Human | interventions — N95 Respirators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N95 Respirator (Active Comparator): Participants in this arm will wear an N95 respirator and safety goggles during Live Attenuated Influenza Vaccine exposure.
  Interventions: Other: N95 Respirator
- Free Air Portable Air Powered Respirator (Experimental): Participants in this arm will wear a Free Air PAPR and safety goggles during Live Attenuated Influenza Vaccine exposure.
  Interventions: Other: Free Air Portable Air Powered Respirator

INTERVENTIONS:
Other: Free Air Portable Air Powered Respirator — The Free Air PAPR is a portable air powered respirator that you will wear like a backpack with a mask and tubing attached.
  Other Names: Free Air PAPR
  Arms: Free Air Portable Air Powered Respirator
Other: N95 Respirator — The N95 respirator is a mask that is standardly used clinically at Wake Forest Baptist Health.
  Arms: N95 Respirator

SUMMARY:
This study will compare the efficacy of the Free Air Portable Air Powered Respirator (PAPR) system versus a N95 mask in preventing nasal detection of influenza following an exposure. The investigators hypothesize the use of the Free Air PAPR system will be superior to a N95 respirator at interrupting the exposure of the study participants to aerosolized influenza virus particles.

DETAILED DESCRIPTION:
Airborne transmission represents one of the most rapidly spreading and least understood dissemination mechanisms for pathogens. Public health strategies to prevent and control the often explosive outbreaks associated with such pathogens are: 1) vaccination and treatment, if available, 2) decontamination of the exposed areas and surfaces, and 3) isolation and barrier precautions such as face masks. Unfortunately, evidence of the efficacy of currently recommended barrier precautions is currently lacking.

Attempts to validate the effectiveness of personal protective equipment are limited to in vitro experiments with mannequin heads. This human exposure study will provide a much more accurate life-like exposure scenario. The use of live attenuated influenza virus vaccine has been proven to be safe.

Objectives: Evaluate the Free Air Portable Air Powered Respirator (PAPR) versus an N95 face mask for preventing the airborne cross-transmission of aerosolized influenza in human participants.

Methods: Participants will be randomized to one of two arms: a) N95 respirator, or b) Free Air PAPR System. The primary outcome will be the rate of the transmission for the 2 study groups, so a nasal and nasopharyngeal swab will be performed immediately following the exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49 years of age
* Employee or student at Wake Forest University School of Medicine and Wake Forest University

Exclusion Criteria:

* Respiratory tract disorders and other chronic diseases, and medical conditions and treatments which are contraindications to mask usage
* Severe claustrophobia or inability to tolerate masks
* Contraindications to FluMist:
* Children younger than 18 years; proposed age range is 18-49
* Adults 50 years and older; proposed age range is 18-49
* People who have received the live attenuated influenza vaccine within 3 weeks of the exposure sessions
* People with a history of severe allergic reaction to any component of the vaccine or to a previous dose of any influenza vaccine
* People who are allergic to eggs
* Pregnant women
* People with weakened immune systems (immunosuppression)
* People who have taken influenza antiviral drugs within the previous 48 hours
* People who care for severely immunocompromised persons who require a protective environment (or otherwise avoid contact with those persons for 7 days after getting the nasal spray vaccine)
* People of any age with asthma might be at increased risk for wheezing after getting the nasal spray vaccine
* The safety of the nasal spray vaccine has not been established in people with underlying medical conditions that place them at high risk of serious flu complications. This includes children and adults who have lung disease, heart disease (except isolated hypertension), kidney disease (like diabetes), kidney or liver disorders, neurologic/neuromuscular, or metabolic disorders. Moderate or severe acute illness with or without fever is a general precaution for vaccination
* Guillain-Barre Syndrome (GBS) within 6 weeks following a previous dose of influenza vaccine is considered a precaution for use of all influenza vaccines
* Treatment with nasal decongestants, nasal antibiotic and/or steroid preparations will not be allowed

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Nasal Swabs | Immediately following Live Attenuated Influenza Vaccine exposure
  A nasal swab will be performed immediately following the exposure.
Nasopharyngeal swabs | Immediately following Live Attenuated Influenza Vaccine exposure
  A nasopharyngeal swab will be performed immediately following the exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Bischoff, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School Of Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Miller MA, Viboud C, Balinska M, Simonsen L. The signature features of influenza pandemics--implications for policy. N Engl J Med. 2009 Jun 18;360(25):2595-8. doi: 10.1056/NEJMp0903906. Epub 2009 May 7. No abstract available. PMID 19423872
- [Background] Institute of Medicine (US) Committee on Personal Protective Equipment for Healthcare Personnel to Prevent Transmission of Pandemic Influenza and Other Viral Respiratory Infections: Current Research Issues; Larson EL, Liverman CT, editors. Preventing Transmission of Pandemic Influenza and Other Viral Respiratory Diseases: Personal Protective Equipment for Healthcare Personnel: Update 2010. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209584/ PMID 24983058
- [Background] Brankston G, Gitterman L, Hirji Z, Lemieux C, Gardam M. Transmission of influenza A in human beings. Lancet Infect Dis. 2007 Apr;7(4):257-65. doi: 10.1016/S1473-3099(07)70029-4. PMID 17376383
- [Background] Bischoff WE, Bassetti S, Bassetti-Wyss BA, Wallis ML, Tucker BK, Reboussin BA, D'Agostino RB Jr, Pfaller MA, Gwaltney JM Jr, Sherertz RJ. Airborne dispersal as a novel transmission route of coagulase-negative staphylococci: interaction between coagulase-negative staphylococci and rhinovirus infection. Infect Control Hosp Epidemiol. 2004 Jun;25(6):504-11. doi: 10.1086/502430. PMID 15242200
- [Background] Bischoff WE, Tucker BK, Wallis ML, Reboussin BA, Pfaller MA, Hayden FG, Sherertz RJ. Preventing the airborne spread of Staphylococcus aureus by persons with the common cold: effect of surgical scrubs, gowns, and masks. Infect Control Hosp Epidemiol. 2007 Oct;28(10):1148-54. doi: 10.1086/520734. Epub 2007 Aug 29. PMID 17828691
- [Background] Gwaltney JM, Hendley JO. Respiratory transmission. In: Epidemiologic methods for the study of infectious diseases. (p.213-227) Thomas JC, Weber DJ (eds). Oxford University Press. 2001, New York, New York.
- [Background] Bischoff WE. Novel Technique to Study Live Influenza and Common Cold Virus in Mono-Dispersed Aerosols. 49th Interscience Conference on Antimicrobial Agents and Chemotherapy. San Francisco, CA, K-1615a, Sept. 12-15, 2009
- [Background] Bischoff WE. Transmission route of rhinovirus type 39 in a monodispersed airborne aerosol. Infect Control Hosp Epidemiol. 2010 Aug;31(8):857-9. doi: 10.1086/655022. PMID 20569111
- [Background] Murayama S, Kawai R, Hirabuki N, Miura T, Mitomo M, Kozuka T, Usio Y. [Intra-arterial ACNU chemotherapy of malignant glioma]. Nihon Igaku Hoshasen Gakkai Zasshi. 1988 Feb 25;48(2):144-53. No abstract available. Japanese. PMID 3164472
- [Background] Bischoff WE, Swett K, Leng I, Peters TR. Exposure to influenza virus aerosols during routine patient care. J Infect Dis. 2013 Apr;207(7):1037-46. doi: 10.1093/infdis/jis773. Epub 2013 Jan 30. PMID 23372182
- [Background] Hayden FG, Albrecht JK, Kaiser DL, Gwaltney JM Jr. Prevention of natural colds by contact prophylaxis with intranasal alpha 2-interferon. N Engl J Med. 1986 Jan 9;314(2):71-5. doi: 10.1056/NEJM198601093140202. PMID 3001519
- [Background] Ford CR, Peterson DE, Mitchell CR. An appraisal of the role of surgical face masks. Am J Surg. 1967 Jun;113(6):787-90. doi: 10.1016/0002-9610(67)90348-0. No abstract available. PMID 6023917
- [Background] Ha'eri GB, Wiley AM. The efficacy of standard surgical face masks: an investigation using "tracer particles". Clin Orthop Relat Res. 1980 May;(148):160-2. PMID 7379387
- [Background] Mitchell NJ, Hunt S. Surgical face masks in modern operating rooms--a costly and unnecessary ritual? J Hosp Infect. 1991 Jul;18(3):239-42. doi: 10.1016/0195-6701(91)90148-2. PMID 1680906
- [Background] Huang C, Willeke K, Qian Y, Grinshpun S, Ulevicius V. Method for measuring the spatial variability of aerosol penetration through respirator filters. Am Ind Hyg Assoc J. 1998 Jul;59(7):461-5. doi: 10.1080/15428119891010208. PMID 9697293
- [Background] Qian Y, Willeke K, Grinshpun SA, Donnelly J, Coffey CC. Performance of N95 respirators: filtration efficiency for airborne microbial and inert particles. Am Ind Hyg Assoc J. 1998 Feb;59(2):128-32. doi: 10.1080/15428119891010389. PMID 9487666
- [Background] Treanor JJ, Kotloff K, Betts RF, Belshe R, Newman F, Iacuzio D, Wittes J, Bryant M. Evaluation of trivalent, live, cold-adapted (CAIV-T) and inactivated (TIV) influenza vaccines in prevention of virus infection and illness following challenge of adults with wild-type influenza A (H1N1), A (H3N2), and B viruses. Vaccine. 1999 Dec 10;18(9-10):899-906. doi: 10.1016/s0264-410x(99)00334-5. PMID 10580204
- [Background] The Rainbow Passage, a public domain text, can be found on page 127 of the 2nd edition of Grant Fairbanks' Voice and Articulation Drillbook. New York: Harper & Row
- See also: American National Standards Institute (ANSI)/ American Society of Heating, Refrigerating and Air-Conditioning Engineers (ASHRAE) 52.2 Method of Testing General Ventilation Air-Cleaning Devices for Removal Efficiency by Particle Size. (Accessed Dec1,2011) — http://webstore.ansi.org/RecordDetail.aspx?sku=ANSI%2FASHRAE%2052.2-2007&source=google&adgroup=ashrae&gclid=CKC5u83K4awCFUqb7Qodcn3FoA